CLINICAL TRIAL: NCT05381337
Title: A Method of Calculating the Shortest Incision for Internal Fixation of Zygomatic Arch Fracture: Sideburns Mini Incision
Brief Title: A Method of Calculating the Shortest Incision for Internal Fixation of Zygomatic Arch Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wei Jing (Other)
Responsible Party: Sponsor-Investigator, Wei Jing, Professor, Sichuan University
Organization: Sichuan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCHSIRB-D-2021-264
Record Dates: First submitted 2022-05-06; First posted 2022-05-19 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Zygomatic Fractures
Keywords: Zygomatic Arch; Fracture Fixation
MeSH Terms: conditions — Zygomatic Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the sideburns mini incision group (Experimental): Forty patients (the sideburns mini incision group) were treated with sideburns mini incision.
  Interventions: Procedure: sideburns mini incision
- the coronal scalp incision group (Other): Forty patients (the coronal scalp incision group) were treated with coronal scalp incision.
  Interventions: Procedure: coronal scalp incision

INTERVENTIONS:
Procedure: sideburns mini incision — The investigators present a new method to calculate the shortest incision for zygomatic fracture, and use this method to calculate the sideburns mini incision for the surgical treatment of zygomatic arch fracture.
  Arms: the sideburns mini incision group
Procedure: coronal scalp incision — Coronal scalp incisions were used as control group.
  Arms: the coronal scalp incision group

SUMMARY:
In this study, a new method was proposed to calculate the length of sideburns mini incision for zygomatic arch fracture. The purpose of this study was to compare the sideburns mini incision calculated by this method with the coronal scalp incision, so as to determine the therapeutic effect and advantages of sideburns mini incision calculated by this method.

DETAILED DESCRIPTION:
Eighty patients with zygomatic arch fracture were treated with surgical intervention. Forty patients were treated with sideburns mini incision, and the other forty patients were treated with coronal scalp incision. Data such as incision length, operation time and postoperative complications were recorded. The follow-up periods were 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and imaging diagnosis of zygomatic arch fracture or zygomatic maxillary complex fracture.
2. Fracture fragments are obviously displaced, which affects the appearance and function of the patient. Simple prying is instable and requires open reduction and internal fixation.
3. No previous surgical treatment.

Exclusion Criteria:

1. Accompanied by multiple fractures of mandible, nasal bone and so on.
2. There are traumatic scars in the operation area, which can be accessed through the original wound.
3. History of bone disease and / or wound healing disorders.
4. Mental and intellectual disorders.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Incision length | during the surgical procedure
  Incision length for open reduction and internal fixation of zygomatic arch fractures.
Operative duration | from the beginning to the end of surgery
  The length of time spent on operation.
Postoperative pain | 24 hours after surgery
  Visual Analogue Scale was used to evaluate the burden of postoperative pain. The maximum score is 10, and the minimum score is 0. Higher scores represent more intense pain.
Postoperative stay | From the end of surgery until discharge, up to 15 days. After evaluation by the same chief knife physician, the patient recovered well postoperatively and could be discharged.
  Days of postoperative hospital stay was calculated to evaluate patient recovery.
Postoperative adverse effects | from the end of surgery to 6 months after surgery
  Including bleeding, malocclusion, infection, nerve injury, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jing, Professor, Study Chair — Department of Oral and Maxillofacial Surgery, West China Hospital of Stomatology, Sichuan University
Locations (1):
- Department of Oral and Maxillofacial Surgery, West China College of Stomatology, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang L, Jiang C, Lin Y, Wen Y, Huang X, Huang J, Lin L. Analysis of Maxillofacial Fractures Based on the Etiology in Southeast China: A 10-Year, Multi-Center Study. J Craniofac Surg. 2021 Jun 1;32(4):1432-1435. doi: 10.1097/SCS.0000000000007183. PMID 33038178
- [Result] Tent PA, Juncar RI, Juncar M. Epidemiological Analysis of Zygomatic Bone Fractures in North-Western Romanian Population: A 10-Year Retrospective Study. In Vivo. 2020 Jul-Aug;34(4):2049-2055. doi: 10.21873/invivo.12006. PMID 32606181
- [Result] Kim JH, Kim YS, Oh DY, Jun YJ, Rhie JW, Moon SH. Efficacy of Altered Two-Point Fixation in Zygomaticomaxillary Complex Fracture. Biomed Res Int. 2020 Mar 18;2020:8537345. doi: 10.1155/2020/8537345. eCollection 2020. PMID 32258152
- [Result] Panneerselvam E, Balasubramanian S, Kempraj J, Babu VR, Raja VBKK. Management of Zygomatic Arch Fractures by Intraoral Open Reduction and Transbuccal Fixation: A Technical Note. Craniomaxillofac Trauma Reconstr. 2020 Jun;13(2):130-132. doi: 10.1177/1943387520911866. Epub 2020 Mar 17. PMID 32642044
- [Result] Cheon JS, Seo BN, Yang JY, Son KM. Clinical Follow-up on Sagittal Fracture at the Temporal Root of the Zygomatic Arch: Does It Need Open Reduction? Arch Plast Surg. 2013 Sep;40(5):546-52. doi: 10.5999/aps.2013.40.5.546. Epub 2013 Sep 13. PMID 24086808
- [Result] Birgfeld CB, Mundinger GS, Gruss JS. Evidence-Based Medicine: Evaluation and Treatment of Zygoma Fractures. Plast Reconstr Surg. 2017 Jan;139(1):168e-180e. doi: 10.1097/PRS.0000000000002852. PMID 28027253
- [Result] Strong EB, Gary C. Management of Zygomaticomaxillary Complex Fractures. Facial Plast Surg Clin North Am. 2017 Nov;25(4):547-562. doi: 10.1016/j.fsc.2017.06.006. PMID 28941507
- [Result] Ling XF, Yew CC, Mohd Nazri SB, Tew MM. Unilateral Zygomatic Complex Fracture - A Comparison Between Nonsurgical Treatment and Surgical Treatment. J Craniofac Surg. 2021 Oct 1;32(7):e627-e630. doi: 10.1097/SCS.0000000000007603. PMID 33654041
- [Result] Sanada Y, Yabuuchi T, Yoshioka H, Kubota H, Kato A. Zigzag skin incision effectively camouflages the scar and alopecia for moyamoya disease: technical note. Neurol Med Chir (Tokyo). 2015;55(3):210-3. doi: 10.2176/nmc.tn.2014-0193. Epub 2015 Feb 20. PMID 25739436
- [Result] Ji SY, Kim SS, Kim MH, Yang WS. Surgical Methods of Zygomaticomaxillary Complex Fracture. Arch Craniofac Surg. 2016 Dec;17(4):206-210. doi: 10.7181/acfs.2016.17.4.206. Epub 2016 Dec 23. PMID 28913285
- [Result] Verpaele A, Tonnard P, Gaia S, Guerao FP, Pirayesh A. The third suture in MACS-lifting: making midface-lifting simple and safe. J Plast Reconstr Aesthet Surg. 2007;60(12):1287-95. doi: 10.1016/j.bjps.2006.12.012. Epub 2007 Jun 29. PMID 17604708
- [Result] Chopan M, Buchanan PJ, Mast BA. The Minimal Access Cranial Suspension Lift. Clin Plast Surg. 2019 Oct;46(4):547-557. doi: 10.1016/j.cps.2019.06.005. Epub 2019 Aug 2. PMID 31514807